CLINICAL TRIAL: NCT02762396
Title: The Norwegian Stroke in the Young Study II
Acronym: NOR-SYSII
Status: Completed | Type: Observational
Sponsor: Haukeland University Hospital (Other)
Collaborators: Helsinki University Central Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2015 / 1769
Record Dates: First submitted 2016-03-01; First posted 2016-05-05 (Estimated); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Ischemic Stroke at a Young Age
Keywords: Young ischemic stroke; Risk factors; Causes; Consequences

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — EDTA-blood and serum will be collected for future analysis
Oversight: Data Monitoring Committee: No

SUMMARY:
NOR-SYS II is designed for finding the cause of acute ischemic stroke lesions in Young adults, age 15 to 49 years. Risk factors, arterial wall changes by intima-media thickness and plaques and consequences of stroke are examined by standardized diagnostics.

DETAILED DESCRIPTION:
NOR-SYS II is as far as possible standardized concerning patients' history, ultrasound examination of pre-cerebral and femoral arteries, and standardized examinations performed by speech therapists, occupational therapists and physiotherapists.

The ultrasound-protocol for carotid and femoral arteries is the same as previously performed in the NOR-SYS study. The Methods have been published before.

ELIGIBILITY:
Inclusion Criteria:

* Documented acute, arterial ischemic stroke
* Speaks Norwegian fluently

Exclusion Criteria:

* Post-traumatic and procedure related stroke
* Sinus venous thrombosis, sepsis and endocarditis
* Serious co-morbidity, such as advanced cancer with "end-of-life stroke".
* Patients mentally retarded or with severe psychiatric disease who do not accept the diagnosis and who would need sedation to perform clinical diagnostics.

Ages: 15 Years to 49 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients with documented ischemic stroke at a young age (< 50 years) in Norway
Sampling Method: Non-Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Established atherosclerosis | Established atherosclerosis will serve as outcome measure for data collected during hospital stay and will be related to risk factors. The data will be presented one year after finishing the 5-years of inclusion of the whole study group.
  The ultrasound protocol of the NOR-SYS study will be applied for carotid and femoral arteries. In addition angiographies will be done for patients with suspicious arterial disease. The measurements will be done within hospital stay after the acute stroke.

SECONDARY OUTCOMES:
New cardiovascular events | One year after the stroke
  Patients With different causes of ischemic stroke have different prognosis that is worst for recurrent stroke and other cardiovascular events for patients with atherosclerosis.
Death | One year after the stroke
  Death fro all causes with subgroups of cardiovascular death, cancer and other causes of death will be registered
Alive but not back to previous education or full-time job | One year after the stroke
  Not back to work because of stroke related problems. Standardized questionnaires will be used to collect information about education and work before stroke and the situation after 3 months and one year. The frequency and reasons why patients did not come back to their education situation or their job they did before the stroke are collected. We expect that it is still possible within a year from stroke onset, to specify the sort of problem related to stroke or unrelated to stroke. This may get more unspecific, the longer the time gets from stroke onset to follow-up. NOR-SYS II will focus on a particular group of patients that seem to function well but that struggle with unvisible problems such as tiredness and reduced capacity / energy to work.

CONTACTS AND LOCATIONS:
Overall Officials: Ulrike Waje-Andreassen, MD, PhD, Principal Investigator — Haukeland University Hospital
Locations (1):
- Dep. of Neurology, Bergen, Norway

IPD SHARING:
Plan to Share IPD: Yes
Contribution to the SECRETO study Contribution to other young ischemic stroke trials, if actual
Supporting Information: Study Protocol
Time Frame: Data can be shared after the study is completed in 2022.
Access Criteria: Actual study protocols have to be approved by the Ethics Committee, and may after approval receive actual data from the NOR-SYS II study

REFERENCES:
- [Background] Fromm A, Thomassen L, Naess H, Meijer R, Eide GE, Krakenes J, Vedeler CA, Gerdts E, Larsen TH, Kuiper KK, Laxdal E, Russell D, Tatlisumak T, Waje-Andreassen U. The Norwegian Stroke in the Young Study (NOR-SYS): rationale and design. BMC Neurol. 2013 Jul 17;13:89. doi: 10.1186/1471-2377-13-89. PMID 23865483